CLINICAL TRIAL: NCT06880627
Title: Brain Boost Program to Improve Cognitive Function in People With Systemic Sclerosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Scleroderma Foundation (Unknown)
Responsible Party: Principal Investigator, Yen T Chen, PhD, Research Assistant Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00267401
Record Dates: First submitted 2025-03-11; First posted 2025-03-18 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Scleroderma
Keywords: Cognitive issues; Memory or Focus problems; Internet connected devices; Online group sessions; Online brain games; Surveys
MeSH Terms: conditions — Scleroderma, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Brain Boost group (Experimental)
  Interventions: Behavioral: Brain Boost group
- Waitlist group (Other)
  Interventions: Other: Waitlist group

INTERVENTIONS:
Behavioral: Brain Boost group — There will be 8 group educational sessions over an 8-week program period to learn strategies for improving cognitive function. Participants will also be asked to engage in 20 minutes, at least 5 times per week online game-like cognitively stimulating activities to improve cognitive health. In addition, surveys will be completed as certain timepoints.
  Arms: Brain Boost group
Other: Waitlist group — This group will continue to receive usual health and care routines. Participants will be asked to complete surveys at certain timepoints that are the same as the boost group. After the 6-month follow-up, participants will receive the intervention materials, which include 8 weekly educational session recordings with slides, 8 weeks' subscription to online brain games, and biweekly online office hours. The office hours, hosted by the principal investigator and a trained patient co-facilitator, will give participants a chance to discuss participant's progress and ask questions.
  Arms: Waitlist group

SUMMARY:
The purpose of this study is to examine whether an 8-week online educational group-based program tailored to people with systemic sclerosis can help improve cognitive function and well-being.

The study team hypothesize that participants that receive the intervention will have better improvements immediately after treatment at week 8 in all cognitive function measures, non-cognitive symptoms, and self-management compared to those in the waitlist control.

ELIGIBILITY:
Inclusion Criteria:

* Have physician-diagnosis of Systemic sclerosis (SSc) (any subtype)
* A score of ≥ 10 on the Perceived Deficits Questionnaire
* A score of ≤ 7 on the 6-Item Cognitive Impairment Test
* Have access to a reliable, internet-connected device (e.g. computer, smartphone, tablet)
* Visual acuity with correction sufficient to work on a computer, smartphone, tablet or screen
* Be able to read, speak, and understand English

Exclusion Criteria:

* Diagnosis of dementia or head injury
* Other neurological disorders that might impact cognition
* Have major psychiatric disorder such as major depression and schizophrenia
* Complex, unstable health issues that would preclude full participation in the study (like a planned surgery or active cancer treatment)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in objective cognitive function from baseline to week 8 | Baseline, 8 weeks
  This will be assessed using the online platform BrainCheck. The following tests will be included: (1) Trail Making A & B (attention and mental flexibility); (2) Stroop Color and Word test (executive function); (3) Digit-Symbol Substitution (processing speed); and (4) Immediate and Delayed Recognition tests (memory). A composite score will be calculated through BrainCheck to assess global cognitive function. The score range is 0-200 a higher score means greater cognitive function.

SECONDARY OUTCOMES:
Change in perceived cognitive function will be measured using the Patient-Reported Outcomes Measurement Information System (PROMIS) cognitive function ability 4a short form | Baseline, 8 weeks
  The PROMIS short form evaluates concentration, sharpness, thinking speed, and memory functioning over the past 7 days on a 5-point Likert scale (1 = not at all to 5 = very much). The scores range from 4-20 with higher score indicating higher cognitive functioning. All PROMIS raw scores will be converted to T-scores, where a higher score indicates a greater degree of the domain assessed.
Change in pain will be measured using the PROMIS pain interference short form | Baseline, 8 weeks
  This is a 4-item short form which assesses pain interference with daily activities, work around the home, social activities, and household chores on a 5-point Likert scale (1 = not at all to 5 = very much). The scores range from 4-20 with higher score indicating higher pain interference. All PROMIS raw scores will be converted to T-scores, where a higher score indicates a greater degree of the domain assessed.
Change in fatigue will be measured using the PROMIS fatigue short form | Baseline, 8 weeks
  This is a 4-items short form which evaluates individuals' fatigue experience and its impact on participant's everyday lives using a 5-point Likert scale (1 = not at all to 5 = very much). The scores range from 4-20 with higher score indicating more fatigue. All PROMIS raw scores will be converted to T-scores, where a higher score indicates a greater degree of the domain assessed.
Change in depressed mood will be measured using the PROMIS depression short form | Baseline, 8 weeks
  This is a 4-item short form which assesses feelings of worthlessness, helplessness, depressed mood, and hopelessness on a 5-point Likert scale (1 = Never to 5 = Always). The scores range from 4-20 with higher score indicating more depressed mood. All PROMIS raw scores will be converted to T-scores, where a higher score indicates a greater degree of the domain assessed.
Change in self-management will be evaluated using the Patient Activation Measure (PAM) | Baseline, 8 weeks
  This is a 13-item measure that assesses patient knowledge, skill, and confidence. Each item is scored from 1 (strongly disagree) to 4 (strongly agree). Scores range from 13 to 52, with higher scores indicating greater confidence and knowledge in patients managing participant's condition.

CONTACTS AND LOCATIONS:
Overall Officials: Yen Chen, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified Individual participant data (IPD) will be shared upon request. The shared dataset will include objective cognitive function data, as well as self-report symptom-related data such as pain, anxiety, depressed mood, sleep disturbance, and perceived self-management improvement. Data will be provided in a format that ensures participant confidentiality and compliance with ethical guidelines.
Supporting Information: Study Protocol
Time Frame: The data will be made available within two year of the study's conclusion and will remain accessible for at least five years.
Access Criteria: Researchers requesting access to the data must submit a formal request detailing the intended use of the dataset. Access will be granted upon approval and execution of a data use agreement that ensures compliance with data confidentiality and ethical research practices.
  At this time, there is no designated online repository for data access. Researchers can request data by contacting the study team at yentchen@med.umich.edu.